CLINICAL TRIAL: NCT04663321
Title: A Phase 2a, Randomized, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of MK-1942 Added to Stable Antidepressant Therapy in Participants With Treatment-Resistant Depression
Brief Title: Efficacy and Safety of MK-1942 When Added to Stable Antidepressant Therapy in Participants With Treatment-Resistant Depression (TRD) (MK-1942-006)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntarily terminated due to benefit/risk assessment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1942-006; MK-1942-006 (Other: MSD)
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-1942 Daily Dose Group (Experimental): Participants receive a total daily dose titrated from 5 mg to 20 mg of MK-1942 twice daily (BID), orally, over 4 weeks of treatment duration: 5 mg in Week 1, 10 mg in Week 2, and 20 mg in Weeks 3 and 4. Participants receive MK-1942 and matching placebo packaged in blister cards with an equal number of capsules administered in the morning and evening regardless of treatment assignment.
  Interventions: Drug: MK-1942; Drug: Placebo
- MK-1942 Intermittent Dose Group (Experimental): Participants receive a total daily dose of 10 mg of MK-1942 twice weekly (BIW), orally, for Weeks 1-4. Participants receive MK-1942 and matching placebo packaged in blister cards with an equal number of capsules administered in the morning and evening regardless of treatment assignment.
  Interventions: Drug: MK-1942; Drug: Placebo
- Placebo (Placebo Comparator): Participants receive a dose-matched placebo BID, orally, for 4 weeks. Participants receive matching placebo packaged in blister cards with an equal number of capsules administered in the morning and evening regardless of treatment assignment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1942 — MK-1942 (5 mg or 10 mg capsules) titrated from 5 mg to 20 mg dose BID or 10 mg BIW over 4 weeks.
  Arms: MK-1942 Daily Dose Group; MK-1942 Intermittent Dose Group
Drug: Placebo — Dose matched placebo capsules BID orally over 4 weeks.

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of daily and intermittent dosing of MK-1942 compared to placebo among participants with Treatment-Resistant Depression (TRD) on a stable course of antidepressant therapy. The dual primary hypotheses of the study are that the daily MK-1942 treatment or intermittent MK-1942 treatment are superior to placebo in reducing Montgomery-Asberg Depression Rating Scale (MADRS) score.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for moderate-to-severe major depressive disorder (MDD) without psychotic features according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria at Visit 1 (Screening)
* Is currently experiencing an episode of moderate-to-severe MDD
* Had an inadequate response to 1 to 4 different courses of antidepressant therapy for the current episode of moderate-to-severe MDD
* Has been on a stable course of antidepressant therapy for ≥4 weeks before Visit 1 (Screening)
* Has not initiated psychotherapy for depressive symptoms in the last 3 months before Visit 1 (Screening) and agrees not to initiate a new psychotherapy for depressive symptoms or to modify their current regimen of psychotherapy for depressive symptoms from Visit 1 (Screening) to Visit 9 (Post-dose Follow-up Visit)
* Male participants are eligible if they agree to the following during the intervention period and for at least 7 days after last dose of study intervention: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or agrees to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* A female participant is eligible to participate if she is not a woman of childbearing potential (WOCBP) or a WOCBP who is not pregnant, breastfeeding, or within 3 months from postpartum. WOCBP should use contraceptive methods that are highly effective as per the study specifications or be abstinent from heterosexual intercourse as their preferred and usual lifestyle, have a negative pregnancy test at screening, immediately prior to the first dosing event, and at regular intervals during the study period, and abstain from breastfeeding during the study intervention period and for at least 7 days after last study intervention
* Has a reliable contact person

Exclusion Criteria:

* Has an ongoing episode of MDD that started more than 2 years before Visit 1 (Screening)
* Has a current or prior history of one or more of the following: a) diagnosis of a psychotic disorder b) chronic convulsive disorder, except febrile seizures during childhood c) neurodegenerative disorder, traumatic brain injury causing ongoing cognitive difficulties, or any chronic organic disease of the central nervous system d) intellectual disability of a severity that would affect the ability of the participant to participate in the study e) bipolar and related disorders, MDD with psychosis f) MDD with mixed features g) posttraumatic stress disorder if not in remission for at least 5 years before Visit 1 (Screening) h) obsessive-compulsive disorder i) autism spectrum disorder
* Meets criteria for substance abuse or dependence disorder currently or within the 12 months before Visit 1 (Screening)
* Has a known allergy or intolerance to the active or inert ingredients in MK-1942
* Has a history of malignancy ≤3 years before Visit 1 (Screening) except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Has a Body Mass Index (BMI) >40 kg/m2
* Has HIV or nonstable hypothyroidism, diabetes, cardiovascular disease, or respiratory disease
* Failed to adequately respond to treatment with ketamine or esketamine for the current or a prior episode of MDD
* Previously received electroconvulsive therapy within the past 10 years, deep brain stimulation, or vagal nerve stimulation for treatment of depression
* Is imminent risk for self harm or harm to others
* Is currently participating in or has previously participated in an interventional clinical study within the 2 months before Visit 1 (Screening), or has participated in >4 interventional clinical studies within the 2 years before Visit 1 (Screening)
* Has known renal disease or is experiencing renal insufficiency
* Routinely consumes >3 alcoholic drinks per day. One standard drink is defined as any beverage containing 14 gram (g) of pure alcohol
* Requires use of a language interpreter to participate in the study
* Had major surgery or donated or lost >1 unit of blood within the 4 weeks before Visit 1 (Screening)
* Is pregnant or is currently breastfeeding or plans to breastfeed during the course of the study
* Is a woman with <12 months of amenorrhea and is receiving hormone replacement therapy (HRT) or an estrogen-based contraceptive
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (45):
- United States (45):
  - University of Alabama at Birmingham - School of Medicine-Psychiatry ( Site 1073), Birmingham, Alabama
  - Preferred Research Partners ( Site 1079), Little Rock, Arkansas
  - Woodland International Research Group ( Site 1017), Little Rock, Arkansas
  - CITrials-Outpatient Facility ( Site 1098), Bellflower, California
  - Axiom Research ( Site 1053), Colton, California
  - Collaborative Neuroscience Network, LLC. ( Site 1032), Garden Grove, California
  - CITrials ( Site 1105), Santa Ana, California
  - Institute of Living ( Site 1061), Hartford, Connecticut
  - Gulfcoast Clinical Research Center ( Site 1110), Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 1116), Hallandale, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare ( Site 1039), Jacksonville, Florida
  - Innovative Clinical Research ( Site 1044), Lauderhill, Florida
  - Behavioral Clinical Research ( Site 1037), Miami, Florida
  - Aqualane Clinical Research ( Site 1113), Naples, Florida
  - APG RESEARCH, LLC ( Site 1087), Orlando, Florida
  - University of South Florida-Psychiatry and Behavioral Neurosciences ( Site 1093), Tampa, Florida
  - K2 Medical Research - Winter Park ( Site 1115), Winter Park, Florida
  - Atlanta Center for Medical Research ( Site 1022), Atlanta, Georgia
  - iResearch Atlanta ( Site 1040), Decatur, Georgia
  - Psych Atlanta ( Site 1108), Marietta, Georgia
  - iResearch Savannah ( Site 1041), Savannah, Georgia
  - Ascension Saint Elizabeth ( Site 1003), Chicago, Illinois
  - CBH Health ( Site 1076), Gaithersburg, Maryland
  - Boston Clinical Trials ( Site 1028), Boston, Massachusetts
  - University of Michigan-Psychiatry ( Site 1051), Ann Arbor, Michigan
  - Altea Research ( Site 1018), Las Vegas, Nevada
  - Hassman Research Institute ( Site 1036), Berlin, New Jersey
  - Global Medical Institutes LLC; Princeton Medical Institute ( Site 1049), Princeton, New Jersey
  - Albuquerque Neuroscience Inc. ( Site 1107), Albuquerque, New Mexico
  - Hapworth Research Inc.-Clinical Research Department ( Site 1090), New York, New York
  - Manhattan Behavioral Medicine ( Site 1096), New York, New York
  - Richmond Behavioral Associates ( Site 1011), Staten Island, New York
  - New Hope Clinical Research ( Site 1082), Charlotte, North Carolina
  - Clinical Trials of America, LLC ( Site 1103), Hickory, North Carolina
  - Neuro-Behavioral Clinical Research ( Site 1045), North Canton, Ohio
  - Paradigm Research Professionals ( Site 1089), Oklahoma City, Oklahoma
  - Suburban Research Associates-Clinical Research ( Site 1042), Media, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System-Mood Disorders Treatment and Research Proga, Philadelphia, Pennsylvania
  - Keystone Clinical Studies ( Site 1031), Plymouth Meeting, Pennsylvania
  - Baylor College of Medicine ( Site 1019), Houston, Texas
  - AIM Trials, LLC ( Site 1111), Plano, Texas
  - Cedar Clinical Research ( Site 1023), Draper, Utah
  - Woodstock Research Center ( Site 1084), Woodstock, Vermont
  - Northwest Clinical Research Center ( Site 1112), Bellevue, Washington
  - Core Clinical Research ( Site 1081), Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and randomized at 27 study sites in the US.
Period: Overall Study
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Started | 40 | 19 | 40
Completed | 28 | 15 | 35
Not Completed | 12 | 4 | 5
Not completed — Study terminated by Sponsor | 2 | 1 | 2
Not completed — Withdrawal by Subject | 10 | 3 | 2
Not completed — Not provided | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo | Total
Number analyzed (Participants) | 40 | 19 | 40 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (12.3) | 48.3 (12.6) | 48.7 (13.3) | 48.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 12 | 26 | 60
  Male | 18 | 7 | 14 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 8 | 12
  Not Hispanic or Latino | 37 | 18 | 32 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 4 | 7 | 22
  White | 27 | 15 | 31 | 73
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to Week 3
Description: The change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) score is presented. MADRS includes 10 participant-rated items, each scored on a scale from 0 (normal, no symptom) to 6 (symptoms of maximum severity) [total scores range from 0 (normal/no symptom) to 60 (severe depression). Higher scores correspond to greater symptom severity, whereas a negative change from baseline score indicates improvement.
Time Frame: Baseline and Week 3
Population: All randomized participants who received ≥1 dose of study intervention, have ≥1 post-treatment and -randomization endpoint observation, and have baseline data available are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 30 | 16 | 37
Units on a scale | -8.1 [-11.5 to -4.6] | -12.5 [-17.3 to -7.7] | -11.4 [-14.6 to -8.1]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.168, ANCOVA; LS Mean Difference = 3.3, 95% CI 2-sided [-1.4 to 8.0]
Statistical Analysis 2: Comparison: MK-1942 Intermittent Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.697, ANCOVA; LS Mean Difference = -1.1, 95% CI 2-sided [-6.9 to 4.7]

2. Primary Outcome: Change From Baseline in MADRS Total Score to Week 1
Description: as for outcome 1
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 37 | 19 | 39
Units on a scale | -5.2 [-7.9 to -2.6] | -6.3 [-10.0 to -2.6] | -8.1 [-10.7 to -5.5]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.124, ANCOVA; LS Mean Difference = 2.9, 95% CI 2-sided [-0.8 to 6.6]
Statistical Analysis 2: Comparison: MK-1942 Intermittent Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.417, ANCOVA; LS Mean Difference = 1.9, 95% CI 2-sided [-2.7 to 6.4]

3. Primary Outcome: Number of Participants Who Experienced An Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 6 Weeks
Population: All randomized participants who received ≥11 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 40 | 19 | 40
Participants | 29 | 13 | 27

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 3
Time Frame: Up to approximately 4 Weeks
Population: All randomized participants who received ≥11 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 40 | 19 | 40
Participants | 4 | 3 | 1

5. Secondary Outcome: Change From Baseline in the Hamilton Depression Rating Scale (HAM-D17) Total Score to Week 3
Description: The HAM-D17 scale was used to evaluate the depressive symptoms experienced over the past week. The HAM-D17 is a 17-item participant-rated scale, with each item scored from 0 to 2 or 4 (depending on the question) reflective of severity (0 is absence of symptom and higher scores indicate greater symptom severity). The total score ranges from 0 (no apparent symptoms) to 52 (most severe symptoms). A negative change from baseline indicates symptom improvement, and vice versa.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 30 | 16 | 37
Units on a scale | -5.5 [-7.7 to -3.3] | -8.2 [-11.2 to -5.1] | -7.5 [-9.6 to -5.5]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.187, ANCOVA; LS Mean Difference = 2.0, 95% CI 2-sided [-1.0 to 5.1]
Statistical Analysis 2: Comparison: MK-1942 Intermittent Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.738, ANCOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-4.3 to 3.1]

6. Secondary Outcome: Change From Baseline in the HAM-D17 Scale Total Score to Week 1
Description: as for outcome 5
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 37 | 19 | 39
Units on a scale | -4.1 [-5.9 to -2.3] | -4.6 [-7.2 to -2.1] | -5.8 [-7.6 to -4.0]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS means; p = 0.182, ANCOVA; LS Mean Difference = 1.7, 95% CI 2-sided [-0.8 to 4.3]

7. Secondary Outcome: Change From Baseline in the Clinician Global Impression-Severity (CGI-S) Total Score to Week 3
Description: The CGI-S is rated on a 7-point scale using a range of responses from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Higher score corresponds to greater symptom severity. A negative change score indicates improvement, and vice versa.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 30 | 16 | 37
Units on a scale | -0.9 [-1.3 to -0.5] | -1.3 [-1.9 to -0.7] | -1.1 [-1.5 to -0.7]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.630, ANCOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 2: Comparison: MK-1942 Intermittent Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.549, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]

8. Secondary Outcome: Change From Baseline in the Clinician Global Impression-Severity (CGI-S) Total Score to Week 1
Description: as for outcome 7
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 37 | 19 | 39
Units on a scale | -0.4 [-0.7 to -0.1] | -0.7 [-1.1 to -0.3] | -0.8 [-1.1 to -0.5]
Statistical Analysis 1: Comparison: MK-1942 Daily Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.062, ANCOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.0 to 0.8]
Statistical Analysis 2: Comparison: MK-1942 Intermittent Dose Group vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.878, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5]

9. Secondary Outcome: Mean Plasma Concentration of MK-1942 Plasma Concentration
Description: The mean plasma concentration of MK-1942 10 mg given as a single or multiple dose regimen was determined.
Time Frame: Day 15: 12 (Daily Dose) or 72 (Intermittent Dose) hours postdose
Population: A subset of MK-1942-treated participants who complied with the protocol sufficiently to ensure that generated data are likely to exhibit the effects of treatment are included.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
Number analyzed (Participants) | 29 | 17 | 0
nM | 130 (69.3) | 9.43 (9.13) |

ADVERSE EVENTS:
Time Frame: Up to ~6 weeks
Description: All treated participants are included.
Arm/Group | MK-1942 Daily Dose Group | MK-1942 Intermittent Dose Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/19 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/19 | 1/40
Other Adverse Events (participants affected / at risk) | 22/40 | 13/19 | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1942 Daily Dose Group (N=40) | MK-1942 Intermittent Dose Group (N=19) | Placebo (N=40)
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1942 Daily Dose Group (N=40) | MK-1942 Intermittent Dose Group (N=19) | Placebo (N=40)
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 6
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
Disease progression (General disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0 | 5
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1
Dizziness (Nervous system disorders) | 10 | 6 | 3
Essential tremor (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 1 | 7
Somnolence (Nervous system disorders) | 1 | 0 | 4
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT04663321/Prot_SAP_000.pdf